CLINICAL TRIAL: NCT02441686
Title: A Phase II Study of the Efficacy and Safety of Lenalidomide, Subcutaneous Bortezomib and Dexamethasone Combination Therapy for Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Phase II Study of Efficacy and Safety of Lenalidomide, Subcutaneous Bortezomib and Dexamethasone Therapy for Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry); Celgene (Industry)
Responsible Party: Principal Investigator, Jacob Laubach, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-508
Record Dates: First submitted 2015-05-08; First posted 2015-05-12 (Estimated); Results first posted 2024-03-04 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Dexamethasone; Calcium Dobesilate; Hematopoietic Stem Cell Mobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide, subcutaneous Bortezomib, Dexamethasone (Experimental): Lenalidomide (R): 25 mg on days 1-14 orally Subcutaneous Bortezomib (sqV): 1.3 mg/m^2 on days 1, 4, 8 and 11 Dexamethasone (d): 20 mg on days 1, 2, 4, 5, 8, 9, 11 and 12 Stem cell mobilization occurs at the end of Cycle 4. Participants may elect to stop treatment at the end of Induction Cycle 4 and proceed to autologous stem cell transplant (ASCT) with melphalan 200 mg/m^2 conditioning, or receive a full 8 cycles of RsqVd induction therapy. RsqVd cycle duration is 21-days.
  Maintenance follows with the specific regimen determined by risk category. High-risk participants defined as those with International Staging System (ISS) stage II or stage III disease and/or high-risk cytogenetics including t(4;14), t(4; 16), del(17p) receive sqV of 1.3 mg/m^2 on days 1 and 15 in addition to R 10mg (15mg after cycle 3 if tolerated) on days 1-21 of 28-day cycle. Standard-risk participants receive R monotherapy.
  Interventions: Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Procedure: Stem Cell Mobilization; Procedure: Autologous Stem Cell Transplant

INTERVENTIONS:
Drug: Bortezomib
  Other Names: Velcade®
Drug: Lenalidomide
  Other Names: Revlimid®
Drug: Dexamethasone
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex
Procedure: Stem Cell Mobilization
Procedure: Autologous Stem Cell Transplant
  Other Names: ASCT

SUMMARY:
This research study is evaluating a combination of three drugs called lenalidomide, subcutaneous (injection under the skin) bortezomib, and dexamethasone (RVD) as a possible treatment for multiple myeloma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational combination of drugs to learn whether the combination of drugs works in treating a specific cancer. "Investigational" means that the combination of drugs is being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved the combination of drugs for your type of cancer.

Each of the individual drugs, lenalidomide , subcutaneous bortezomib, and dexamethasone, are approved by the U.S. Food and Drug Administration (FDA). The combination has not been approved yet for multiple myeloma or any other type of cancer. Subcutaneous bortezomib is currently approved by the U.S. FDA for the treatment of patients with relapsed/refractory multiple myeloma. Lenalidomide is currently approved for use with dexamethasone for patients with multiple myeloma who have received at least one prior therapy and for the treatment of certain types of myelodysplastic syndrome (another form of cancer affecting the blood). Both Bortezomib and Lenalidomide kill tumor cells and help the body cells to fight cancer. Dexamethasone is commonly used, either alone, or in combination with other drugs, to treat multiple myeloma. Dexamethasone heps to reduce irritation and cell injury (inflammation).

In this research study, the investigators are looking to explore the drug combination of lenalidomide, subcutaneous bortezomib and dexamethasone to see what side effects it may have and how well it works for treatment of newly diagnosed multiple myeloma. This 3 drug regimen showed promising results in previous studies, however administration of intravenous bortezomib caused high levels of nerve injury (a condition involving the nerves of the upper and lower extremities associated with numbness, tingling and burning). In this study, the investigators are testing the hypothesis that subcutaneous administration of bortezomib will result in less nerve toxicity. Therefore, the combination of lenalidomide, dexamethasone and subcutaneous bortezomib may be better tolerated and may allow for a longer duration of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic MM, according to International Myeloma Foundation 2003 Diagnostic Criteria:

  * Clonal plasma cells >10% on bone marrow biopsy
  * A monoclonal protein (paraprotein) in either serum or urine(except in cases of non-secretory myeloma)*
  * Myeloma-related organ dysfunction (1 or more) of the following (evidence of end-organ damage felt related to the plasma cell disorder related organ or tissue impairment (ROTI), commonly referred to by the acronym "CRAB"):

    * Serum Ca ≥ 10.5 mg/dL or
    * Renal insufficiency attributable to myeloma. Serum creatinine > 2mg/dL
    * Anemia: Normochromic, normocytic with a hemoglobin value > 2g/dL below the lower limit of normal or a hemoglobin <10 g/dL
    * Bone lesions (lytic lesions, severe osteopenia or pathologic fractures) or osteoporosis. *If no monoclonal protein is detected (non-secretory disease), then >/= 30% monoclonal bone marrow plasma cells and/or a biopsy-proven plasmacytoma required.
* Has received no prior treatment with any systemic therapy for the treatment of multiple myeloma

  * Prior treatment of hypercalcemia or spinal cord compression with corticosteroids does not disqualify the patient (the dose should not exceed the equivalent of 160 mg of dexamethasone in a 2 week period).
  * Bisphosphonates are permitted.
  * Local radiation as long as two weeks have lapsed since last date of radiotherapy, which is recommended to be a limited field.
* Age ≥18 years at the time of signing Informed Consent
* ECOG performance status ≤ 2 (Karnofsky ≥ 50%)
* Voluntary written informed consent
* Subject must be able to adhere to the study visit schedule and other protocol requirements.

  * Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 µL/mL 10 to14 days prior to therapy and repeated again within 24 hours prior to prescribing lenalidomide for Cycle 1 and must either commit to complete abstinence from heterosexual contact or begin TWO acceptable methods of birth control, one highly effective method and one additional effective (barrier) method, AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must practice complete abstinence or agree to use a condom during sexual contact with a FCBP even if they have had a successful vasectomy. All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program- Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Renal insufficiency (serum creatinine levels > 2.5 mg/dL, calculated Crcl with Cockcroft-Gault formula, see Appendix B, < 45 ml/min)
* Subjects with evidence of mucosal or internal bleeding and/or platelet refractory (i.e., unable to maintain a platelet count ≥ 50,000 cells/mm3)
* Subjects with an absolute neutrophil count (ANC) < 1000 cells/mm3. Growth factors may not be used to meet ANC eligibility criteria
* Subjects with a hemoglobin < 8.0 g/dL
* AST (SGOT) and ALT (SGPT) > 2 x institutional ULN, bilirubin levels ≥1.5 institutional ULN
* Concomitant therapy medications that include corticosteroids (except as indicated in inclusion criteria).
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (Appendix C), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Clinically relevant active infection requiring treatment (antibiotics, antivirals, antifungals).
* Any serious co-morbid condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study.
* Female subject is pregnant or breast-feeding.
* Serious psychiatric illness or addiction likely to interfere with participation in this clinical study.
* Uncontrolled diabetes mellitus.
* Contraindication to any required concomitant drugs or supportive therapies including hypersensitivity to all anticoagulation and antiplatelet options or hypersensitivity to acyclovir or similar anti-viral drug.
* History of allergic reaction/hypersensitivity attributed to compounds containing boron, mannitol, polysorbate 80 or sodium citrate dehydrate.
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes).
* Known seropositive for or active HIV infection or hepatitis B or C viral infection.

  * Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Known intolerance to steroid therapy.
* Patient has hypersensitivity to bortezomib, boron, or mannitol.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Radiation therapy within 2 weeks of enrollment. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 2 weeks have elapsed since the last date of therapy.
* Participant must be able to swallow pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2025-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Laubach, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Eastern Maine Medical Center, Brewer, Maine
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Virginia Piper Cancer Institute, Coon Rapids, Minnesota
  - Virgina Piper Cancer Institute, Minneapolis, Minnesota
  - Hematology Oncology of Northern New Jersey, Morristown, New Jersey

REFERENCES:
- [Result] O'Gorman P, Laubach JP, O'Dwyer ME, Krawczyk J, Yee AJ, Gilligan O, Cahill MR, Rosenblatt J, Quinn J, Murphy PT, DiPietro H, Perera MR, Crotty GM, Cummings K, Hayden PJ, Browne P, Savell A, O'Leary HM, O'Keeffe D, Masone K, Hennessy BJ, Guerrero Garcia T, Scott K, Saeed K, Bianchi G, Dowling P, Tierney C, Richardson PG. Phase 2 studies of lenalidomide, subcutaneous bortezomib, and dexamethasone as induction therapy in patients with newly diagnosed multiple myeloma. Am J Hematol. 2022 May;97(5):562-573. doi: 10.1002/ajh.26491. Epub 2022 Feb 18. PMID 35132679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from December 2015 to June 2017.
Period: Induction
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Started | 46
Safety | 42
Progression-free Survival Evaluable | 41
Evaluable for Induction Response | 40
Received Autologous Stem Cell Transplant (ASCT) | 15
Completed | 38
Not Completed | 8
Not completed — Adverse Event | 4
Not completed — Complicating disease | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Did not receive treatment | 1
Period: Maintenance
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Started | 38
Safety | 35
Completed (Given treatment duration is not a fixed duration, all participants are considered as 'Not Completed'. Reasons off-treatment are provided for all participants not still on treatment as of the date of data extraction.) | 0
Not Completed | 38
Not completed — Remaining on Treatment | 23
Not completed — Physician Decision | 1
Not completed — Adverse Event | 3
Not completed — Progressive Disease | 10
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The analysis population is all enrolled participants.
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 61.5 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2
ECOG Performance Score (PS) [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) PS: (PS0) Fully active, able to carry on all pre-disease performance without restriction (PS1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (PS2) Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about >50% of waking hours
  participants
    ECOG PS 0 | 19
    ECOG PS 1 | 21
    ECOG PS 2 | 2
    Unknown | 4

OUTCOME MEASURES:

1. Primary Outcome: 4-Cycle Induction Overall Response Rate (ORR)
Description: 4-cycle ORR was defined as the percentage of participants who achieved partial response or better based on the International Myeloma Working Group Response (IMWG) criteria during the first 4 cycles of induction therapy.
Time Frame: Participants were followed up to 12 weeks.
Population: Evaluable for disease response analysis having started therapy and assessed for disease post-baseline.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 40
percentage of participants | 95 [85 to 99]

2. Primary Outcome: Induction Overall Response Rate (ORR)
Description: Induction ORR was defined as the percentage of participants who achieved partial response or better based on the International Myeloma Working Group Response (IMWG) criteria during induction therapy either 4 cycles or 8 cycles of combination therapy. Response on ASCT is not included.
Time Frame: Participants were followed up to 24 weeks.
Population: Evaluable for disease response analysis having started therapy and assessed for disease post-baseline.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 40
percentage of participants | 97.5 [89 to 99]

3. Primary Outcome: Four-cycle Induction Peripheral Neuropathy (PN) Rate
Description: Four-cycle induction PN rate was defined as the proportion of participants who experienced peripheral neuropathy includes any attribution and any grades based on the Common Toxicity Criteria for Adverse Events Version 4.0 (CTCAEv4) during the first 4 cycles of induction therapy.
Time Frame: Participants were followed up to 12 weeks.
Population: Safety- all treated population.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 42
proportion of participants | 0.71 [0.58 to 0.83]

4. Primary Outcome: Grade 3-4 Induction Peripheral Neuropathy Rate
Description: Grade 3-4 induction peripheral neuropathy rate was defined as the proportion of participants who experienced grade 3 or 4 peripheral neuropathy based on the Common Toxicity Criteria for Adverse Events Version 4.0 (CTCAEv4) as reported on case report forms during induction therapy (4 cycles RsqVd for ASCT patients and 8 cycles for non-ASCT patients).
Time Frame: Participants were followed up to 24 weeks.
Population: The analysis population is comprised of all treated participants.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 42
proportion of participants | 0.07 [0.02 to 0.17]

5. Secondary Outcome: Median Time to Progression (TTP)
Description: Median TTP based on KM method is defined as the time from first dose of treatment to the first progression event or censored at date last disease assessment. PD, based on IMWG criteria, requires 1+ of the following: >25% increase in the level of serum monoclonal paraprotein, which must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation. >25% increase in 24h urinary light chain excretion, which must also be an absolute increase of at least 200 mg/24 h and confirmed on a repeat investigation. >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10%. Definite increase in the size of existing lytic bone lesions or soft tissue plasmacytomas. Development of new bone lesions or soft tissue plasmacytomas. Development of hypercalcemia.
Time Frame: Disease was assessed up to 41.2 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 41
Months | NA [29.7 to NA] — Limited number of participants progressed during the observation period.

6. Secondary Outcome: 1-Year Progression Free Survival (PFS) Probability
Description: 1-year PFS is the probability estimate at 1 year based on the Kaplan-Meier method. PFS is defined as the duration of time from study entry to documented disease progression or death from any cause, censored at the date last known progression-free for those who have not progressed or died. PD, based on IMWG criteria, requires 1+ of the following: >25% increase in the level of serum monoclonal paraprotein, which must also be an absolute increase of at least 5 g/L and confirmed on a repeat investigation. >25% increase in 24h urinary light chain excretion, which must also be an absolute increase of at least 200 mg/24 h and confirmed on a repeat investigation. >25% increase in plasma cells in a bone marrow aspirate or on trephine biopsy, which must also be an absolute increase of at least 10%. Definite increase in the size of existing lytic bone lesions or soft tissue plasmacytomas. Development of new bone lesions or soft tissue plasmacytomas. Development of hypercalcemia.
Time Frame: Median follow up for PFS is 13.4 months with the relevant observation timepoint equal to 1 year.
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 41
percentage probability | 89.2 [79.2 to 99.3]

7. Secondary Outcome: Median Duration of Response (DOR)
Description: DOR was defined at the time from the first assessment indicating PR or better response to the first progression (PD) event based on IMWG criteria.
Time Frame: Disease was assessed up to 41.2 months.
Population: The analysis population is comprised of participants who achieved partial response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 40
Months | NA [24.2 to NA] — The data are not mature because follow-up for events is not long enough. As such, the median was not reached and the upper bound 95% CI could not be estimated.

8. Secondary Outcome: 1-year Overall Survival (OS) Rate
Description: 1-year OS rate was defined as the percentage of participants alive at 1 year.
Time Frame: Survival was assessed up to 1 year.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone
Number analyzed (Participants) | 42
percentage of participants | 100 [93 to 100]

ADVERSE EVENTS:
Time Frame: AEs were assessed for a maximum of 274 days on induction +30 days, 1071 days on maintenance +30 days.
Description: The analysis population is comprised of all treated participants both starting induction and starting maintenance. SAEs are defined per protocol and OAEs represent all remaining adverse events collected (any treatment attribution and any grade) reported on study case report forms. SAEs and OAEs are reported as maximum grade by toxicity type.
Groups:
- Lenalidomide, Subcutaneous Bortezomib, Dexamethasone - Induction Phase: Lenalidomide (R): 25 mg on days 1-14 orally Subcutaneous Bortezomib (sqV): 1.3 mg/m^2 on days 1, 4, 8 and 11 Dexamethasone (d): 20 mg on days 1, 2, 4, 5, 8, 9, 11 and 12 Stem cell mobilization occurs at the end of Cycle 4. Participants may elect to stop treatment at the end of Induction Cycle 4 and proceed to autologous stem cell transplant (ASCT) with melphalan 200 mg/m^2 conditioning, or receive a full 8 cycles of RsqVd induction therapy. RsqVd cycle duration is 21-days.
- Lenalidomide, [Subcutaneous Bortezomib] - Maintenance Phase: Maintenance follows induction with the specific regimen determined by risk category. High-risk participants defined as those with International Staging System (ISS) stage II or stage III disease and/or high-risk cytogenetics including t(4;14), t(4; 16), del(17p) receive sqV of 1.3 mg/m^2 on days 1 and 15 in addition to R 10mg (15mg after cycle 3 if tolerated) on days 1-21 of 28-day cycle. Standard-risk participants receive R monotherapy.
Arm/Group | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone - Induction Phase | Lenalidomide, [Subcutaneous Bortezomib] - Maintenance Phase
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/35
Serious Adverse Events (participants affected / at risk) | 8/42 | 8/35
Other Adverse Events (participants affected / at risk) | 42/42 | 30/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone - Induction Phase (N=42) | Lenalidomide, [Subcutaneous Bortezomib] - Maintenance Phase (N=35)
Retinal vascular disorder (Eye disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Mania (Psychiatric disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Subcutaneous Bortezomib, Dexamethasone - Induction Phase (N=42) | Lenalidomide, [Subcutaneous Bortezomib] - Maintenance Phase (N=35)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Acoustic nerve disorder NOS (Nervous system disorders) | 1 | 0
Alkaline phosphatase increased (Investigations) | 3 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Anemia (Blood and lymphatic system disorders) | 11 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 1
Anxiety (Psychiatric disorders) | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 9
Bacteraemia (Infections and infestations) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 2
Blurred vision (Eye disorders) | 7 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 3 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac arrthymia (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Chills (General disorders) | 1 | 5
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Cognitive disorder (Psychiatric disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Cold sweat (General disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 2 | 0
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 23 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Creatinine increased (Investigations) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 11 | 12
Dizziness (Nervous system disorders) | 10 | 2
Dry eye (Eye disorders) | 2 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2
Dysesthesia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 8 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Ear pain (Ear and labyrinth disorders) | 1 | 0
Edema face (General disorders) | 2 | 0
Edema limbs (General disorders) | 16 | 7
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 1
Erythema (Eye disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
External ear pain (Ear and labyrinth disorders) | 1 | 0
Eye discharge (Eye disorders) | 0 | 1
Eye infection (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Eye oedema (Eye disorders) | 1 | 0
Eyelid infection (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1
Fatigue (General disorders) | 24 | 9
Fever (General disorders) | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Flatulence (Gastrointestinal disorders) | 1 | 1
Flu like symptoms (General disorders) | 0 | 2
Flushing (Vascular disorders) | 2 | 0
Folliculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal infection (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 | 0
GGT increased (Investigations) | 3 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Gout (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 11 | 2
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hepatitis viral (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hot flashes (Vascular disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyperchloraemia (Investigations) | 0 | 1
Hypercholesterolaemia (Investigations) | 23 | 11
Hyperglycemia (Metabolism and nutrition disorders) | 14 | 11
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphatemia (Investigations) | 1 | 0
Hypertension (Vascular disorders) | 7 | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14 | 8
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypocholesterolaemia (Investigations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 5 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 6
Hypotension (Vascular disorders) | 3 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 2
Injection site erythema (General disorders) | 1 | 0
Injection site erythema (Skin and subcutaneous tissue disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 13 | 5
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Malaise (General disorders) | 3 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0
Mood swings (Nervous system disorders) | 1 | 0
Movements involuntary (Nervous system disorders) | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 4 | 0
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 8
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neuropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 16 | 18
Non-cardiac chest pain (General disorders) | 1 | 0
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 10 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 8
Palpitations (Cardiac disorders) | 1 | 1
Papulopustular rash (Infections and infestations) | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 33 | 11
Personality change (Psychiatric disorders) | 6 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Platelet count decreased (Investigations) | 6 | 6
Pneumonia (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 3
Rectal pain (Gastrointestinal disorders) | 1 | 0
Renal impairment (Investigations) | 1 | 0
Restlessness (Psychiatric disorders) | 2 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 3 | 1
Sinusitis (Infections and infestations) | 2 | 1
Skin infection (Infections and infestations) | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Steroid diabetes (Endocrine disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Taste disorder (Nervous system disorders) | 4 | 0
Temperature regulation disorder (General disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 3
Tongue blistering (General disorders) | 1 | 0
Tooth disorder (Nervous system disorders) | 1 | 0
Transaminitis (Investigations) | 13 | 7
Tremor (Nervous system disorders) | 5 | 0
Upper respiratory infection (Infections and infestations) | 16 | 14
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract discomfort (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Visual disorder (Eye disorders) | 1 | 1
Vitreous hemorrhage (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 4
Weakness in right arm (Nervous system disorders) | 1 | 0
Weight gain (Investigations) | 5 | 0
Weight loss (Investigations) | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
White blood cell decreased (Investigations) | 5 | 6
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT02441686/Prot_SAP_000.pdf